CLINICAL TRIAL: NCT02178189
Title: Randomized Clinical Trial of High vs. Standard-Calorie Formula for Methadone-Exposed Infants
Brief Title: RCT of High- vs. Standard-Calorie Formula for Methadone-Exposed Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Debra L. Bogen, Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO09120457; R21DA029257 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: prenatal opioid exposure; infant; weight gain; infant formula
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Weight Gain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-calorie infant formula (Active Comparator): Infants assigned to this arm were fed standard-calorie infant formula (20 kcal/oz) from 72 hours of life until 21 days of age.
  Interventions: Other: Standard Calorie Infant Formula
- High-calorie infant formula (Experimental): Infants assigned to this arm were fed high-calorie infant formula (24 kcal/oz) from 72 hours of life until 21 days of age.
  Interventions: Other: High Calorie Infant formula

INTERVENTIONS:
Other: High Calorie Infant formula — Infants were randomized to be fed high calorie formula from 72 hours of life until age 21 days.
  Arms: High-calorie infant formula
Other: Standard Calorie Infant Formula — Infants were randomized to be fed standard calorie formula from 72 hours of life until age 21 days.
  Arms: Standard-calorie infant formula

SUMMARY:
Neonatal abstinence syndrome (NAS) symptoms contribute to poor infant weight gain. Early caloric enhancement for infants exposed to methadone is inexpensive, readily available, easy to implement and could improve early outcomes for these high-risk infants. We will conduct a preliminary randomized clinical trial of high-calorie vs. standard-calorie formula for methadone exposed infants to evaluate the adequacy of recruitment, protocol feasibility and estimates of whether high-calorie formula results in more normal patterns of weight loss and gain, less severe NAS symptoms and shorter hospital stays.

DETAILED DESCRIPTION:
Background: Infants exposed to methadone during pregnancy experience high rates of neonatal abstinence syndrome (NAS). Common NAS symptoms (tremulousness, increased muscle tone, sweating, excessive crying, vomiting and diarrhea) increase infants' metabolic needs. Another frequent NAS symptom, weak and uncoordinated suckling, impairs infants' ability to take in adequate calories. These combined problems compromise infant weight gain. The current standard of care for opiate-exposed infants requires evidence of poor weight gain or excessive weight loss before initiating high-calorie formula. We hypothesize that inadequate caloric intake among methadone exposed infants may result in excessive weight loss, slow weight regain and exacerbation of NAS. These factors lead to the newborn's requirement for higher morphine doses and longer duration of hospitalization. Therefore, methadone exposed infants may benefit from early caloric enhancement. A nutritional intervention for opiate-exposed infants has not been previously evaluated. This application will provide data on adequacy of recruitment, protocol feasibility, performance of selected measures, and preliminary estimates of efficacy for a comprehensive R01 submission.

Specific Aims:

1. For methadone exposed infants, compare infants randomized to high (24 kcal/oz) versus standard (20 kcal/oz) formula for the following outcomes:

   * Weight loss and gain patterns. The primary dependent measure will be days until the infant returns to birth weight. Secondary measures will be maximum percent weight loss and days to weight nadir.
   * NAS severity measured by: a) total length of hospital stay for NAS; b) duration of NAS treatment; c) mean Finnegan scores on days 2-10; d) maximum concentration of morphine used to treat NAS.
2. Describe the suck quality at 4-6 days of age among methadone exposed infants. Evaluate the association between the infant suck quality and infant weight loss and gain patterns and measures of NAS severity.

Design: Women on methadone will be recruited during pregnancy and will attend a single brief visit late in pregnancy. After delivery, infants will be randomized in a double blind trial of either high-calorie or standard-calorie formula which will be started at 72 hours after birth and be continued through 21 days of age. Infants will be weighed daily and will have outpatient study visits at 1 and 3 months. For this pilot study, up to 70 mothers will be enrolled over 18 months. This pilot study is needed to establish the feasibility of the study methods and to better estimate differences that can be observed between the groups. For the primary outcome variable, days until the infant returns to birth weight, discrete survival methods will be used.

Potential Impact: Early caloric enhancement for methadone-exposed infants is inexpensive, readily available, easy to implement and could improve outcomes of these high-risk infants. High-calorie formula could result in a more normal pattern of weight loss and gain, less severe NAS symptoms and shorter hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Infants born to pregnant women, who are 18 to 45 years of age, participating in a licensed methadone maintenance treatment program
* planning to delivered at Magee if consented during pregnancy or delivered at Magee within the past 48 hours

Exclusion Criteria:

* Infants born weighing <2200 grams or before 35 weeks
* Multiple gestation pregnancies (eg. twins)
* Infants with major congenital malformations that could interfere with feeding or weight gain, such as Downs syndrome, cleft lip or palate, congenital heart disease or cystic fibrosis will be excluded.
* Infants admitted to the NICU longer than 48 hours for a medical condition other than treatment of NAS
* Women who do not speak English will be excluded because study staff will not be able to communicate effectively.
* Women who intend to place their infant for adoption
* Women who plan on feeding their baby soy formula from birth

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Weight Patterns (gain and loss) | Up to 3 weeks
  Weight loss and gain patterns will include days to return to birth weight, days to weight nadir (lowest point) and maximum percent weight loss.

SECONDARY OUTCOMES:
Neonatal abstinence syndrome (NAS) severity measures | Up to 3 weeks
  NAS (Neonatal abstinence syndrome) severity can be measured in a few ways - for this study, we will use total length of hospital stay for NAS, duration of NAS treatment, mean Finnegan scores on days 3-10 and maximum concentration of morphine used to treat NAS

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Bogen, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States